CLINICAL TRIAL: NCT00557739
Title: A Single-Center, Randomized, Double-Blind, Vehicle-Controlled Study to Assess the Activity of CRx-191 in Reducing the Psoriatic Infiltrate Band Thickness in Plaque Psoriasis
Brief Title: Study of CRx-191 to Assess Activity in Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zalicus (Industry)
Collaborators: Bioskin GmbH (Industry)
Responsible Party: Medical Monitor, CombinatoRx
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRx-191-001; Eudra CT #: 2006-005848-87
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2007-12

CONDITIONS: Plaque Psoriasis
Keywords: CRx-191; Plaque; Psoriasis; nortriptyline hydrochloride; mometasone furoate; psoriatic infiltrate
MeSH Terms: conditions — Plaque, Amyloid; Psoriasis | interventions — Mometasone Furoate; Nortriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): CRx-191 (0.1% mometasone furoate + 0.05% nortriptyline HCl)
  Interventions: Drug: mometasone furoate; Drug: nortriptyline HCl
- 2 (Experimental): CRx-191 (0.1% mometasone furoate + 0.1% nortriptyline HCl)
  Interventions: Drug: mometasone furoate; Drug: nortriptyline HCl
- 3 (Active Comparator): 0.1% mometasone furoate
  Interventions: Drug: mometasone furoate
- 4 (Active Comparator): 0.05% nortriptyline HCl
  Interventions: Drug: nortriptyline HCl
- 5 (Active Comparator): 0.1% nortriptyline HCl
  Interventions: Drug: nortriptyline HCl
- 6 (Placebo Comparator): Vehicle (placebo)
  Interventions: Drug: Vehicle (placebo)

INTERVENTIONS:
Drug: mometasone furoate — Topical 0.1% mometasone furoate
  Arms: 1; 2; 3
Drug: nortriptyline HCl — Topical 0.05% or 0.1% nortriptyline HCl
  Arms: 1; 2; 4; 5
Drug: Vehicle (placebo) — Topical placebo
  Arms: 6

SUMMARY:
CRx-191 is a proprietary synergistic combination drug candidate being evaluated by CombinatoRx for topical psoriasis therapy. CRx-191 was identified via a proprietary screening assay for novel drug combinations demonstrating enhanced inhibition of tumor necrosis factor- alpha and interferon-gamma release, cytokines that are implicated in the pathogenesis of psoriasis.

This clinical trial will assess the effectiveness of CRx-191 in reducing the psoriatic infiltrate band thickness as measured by transdermal ultrasound. All subjects will receive all treatments in separate test fields, with intra-individual comparison of the treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily give written informed consent
* Subject must be between 18 and 70 years of age
* Subject must have chronic plaque psoriasis and stable plaques in an area sufficient for six treatment fields
* The physical examination must be without disease findings unless the investigator considers an abnormality to be irrelevant to the outcome of the study
* Sexually active females of childbearing potential should either be surgically sterile (hysterectomy or tubal ligation), or should use a highly effective medically accepted contraceptive regimen

Exclusion Criteria:

* Erythrodermic, guttate or pustular psoriasis
* Cardiac disease, including recent myocardial infarction, any degree of heart block or other cardiac arrhythmias and valvular heart disease
* Mania
* Narrow angle glaucoma
* Hyperthyroidism by medical history, thyroid stimulating hormone (TSH) less than lower limit of normal (LLN), or receiving thyroid medication
* Intolerance to Lidocaine
* Severe liver disease (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) laboratory values that exceed 1.5x upper limit of normal (ULN))
* Inflammatory dermatoses except psoriasis; bacterial, viral and fungal skin infections; facial rosacea
* Active varicella, tuberculosis, syphilis or post-vaccine reaction
* Autoimmune disease other than plaque psoriasis (e.g. lupus erythematosis and psoriatic arthritis)
* Known allergic reactions or hypersensitivity to any of the components of the study preparations
* Allergy to adhesives on the hydrocolloid dressing used in this study
* UV therapy in the four weeks before the study
* History of malignancy (except for treated or excised basal cell carcinoma)
* Surgery within the previous 3 months (except for minor cosmetic or dental procedures)
* History of drug or alcohol abuse (as defined by the Investigator)
* Symptoms of a clinically significant illness in the four weeks before the study that may influence the outcome of the study
* Positive for HIV antibody
* Subjects who require systemically acting medications for the treatment of psoriasis which might counter or influence the study objectives such as: Methotrexate; Cyclosporine; Anti-TNFα therapies
* Subjects who require medications that inhibit the CYP450 2D6 pathway such as: Quinidine; Cimetidine; Type 1 antiarrhythmics; Phenothiazines; Selective serotonin reuptake inhibitors such as fluoxetine, paroxetine, and sertraline; Reserpine, other anticholinergic drugs, and sympathomimetic drugs
* Topical treatments for psoriasis (except for salicylic acid in vaseline) in the four weeks preceding and during the study (topical corticosteroids disallowed for eight weeks prior to the study)
* Systemic treatments in the two weeks preceding and during the study that may interact with any of the study drugs, such as: Glucocorticoids (po, im, iv); MAO inhibitors; Anti-depressants; Anti-seizure medications; Anti-psychotics; Antihistamines
* Treatments in the two weeks preceding and during the study that may aggravate psoriasis, such as: Anti-malarials; Beta-blockers
* Participation in another clinical trial and/or treatment received with any investigational agent within one month before the initial dose of study medication
* Female subject who is pregnant or lactating
* Significant UV exposure in the four weeks before the study
* Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's return for follow-up visits on schedule
* Other unspecified reasons that, in the opinion of the Investigator or sponsor make the subject unsuitable for enrollment
* Subject is institutionalized because of legal or regulatory order

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the difference in reduction from baseline in psoriatic infiltrate at Day 12 between CRx-191 and vehicle. | Day 12

SECONDARY OUTCOMES:
Differences in reduction from baseline in psoriatic infiltrate at Day 12 between CRx-191 and its components, mometasone furoate and nortriptyline HCI. Demonstrate tolerability and safety of CRx-191. | Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Gassmueller, M.D., Principal Investigator — Bioskin GmbH
Locations (1):
- bioskin GmbH, Berlin, Germany